CLINICAL TRIAL: NCT03333460
Title: Cracking Addiction: Does BRAIN Stimulation-induced Neuroplasticity Reverse Prefrontal Cortex Hypoactivity in Cocaine and neW stImulanTs addiCtion in Humans? (BRAIN SWITCH)
Brief Title: Transcranial Magnetic Stimulation for Cocaine Addiction
Acronym: BRAINSWITCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Giovanni Martinotti, Researcher, ITAB - Institute for Advanced Biomedical Technologies
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: v.1_8/05/2017
Record Dates: First submitted 2017-09-21; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Cocaine Dependence; Substance Use Disorders; Chemical Addiction; Mental Disorder; Cocaine-Related Disorders; Drug Dependence
Keywords: cocaine; addiction; transcranial magnetic stimulation; neuromodulation; neuroimaging; brain stimulation
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Mental Disorders; Behavior, Addictive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: double blind, randomized, sham-controlled with a 1:1 allocation into 2 parallel arms
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: With regard to the treatment, to ensure that both participants and investigators are blind to the condition (active or sham), the selection of the operation mode (15 Hz, sham) will be pre-programmed by member of the that will not be involved in data collection and analysis. Study personnel will not know which mode is being activated. Sham stimulation will use the same coil placement as that used for active stimulation. Outcomes Assessors will not be present during the rTMS sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Active rTMS (15 Hz) (Experimental): The intervention will be Repetitive Transcranial Magnetic Stimulation. Each patient will receive active stimulation targeting the left dorsolateral prefrontal cortex (lDLPFC) with a frequency of 15 Hz and 100% of the individual resting motor threshold, for a total of 40 trains (60 stimuli per train, inter-train interval of 15 second, total duration 13 minutes). Each session will be repeated twice/daily for 10 consecutive days for 2 weeks, during the continued treatment phase. Following this, the participants will receive the maintenance intervention of 2 sessions per week for 3 months (rTMS follow-up), at the same parameters described above. Device: MagPro R30 with the Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham Comparator: Sham rTMS (15 Hz) (Placebo Comparator): The intervention will be Repetitive Transcranial Magnetic Stimulation (Sham). rTMS will be used with the software necessary for the operator to remain blind to the stimulation condition. Also, the software will be pre-programmed by a staff member that will not be involved in data collection and analysis. The sham condition will match the number of pulses delivered during the 15Hz session and will use the same coil placement but the intensity of stimulation will be set a 3% of the individual resting motor threshold so to ensure that the participant will feel similar scalp sensations experienced by participants receiving active rTMS, but brain tissue will not be stimulated. Device: MagPro R30 with the Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS is a non-invasive brain stimulation technique. The investigators will use a MagPro R30 with the Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Other Names: rTMS

SUMMARY:
Background: Cocaine use disorders (CUD) is a complex brain disorder, involving several brain areas and neurocircuits. Effective treatments for CUD are still needed. Repetitive transcranial magnetic stimulation (rTMS) stimulates non-invasively parts of the brain. Preliminary data suggest that rTMS may help reducing cocaine craving and consumption. Researchers want to learn how the brain and the drug-seeking behavior may change with this treatment.

Objectives: To test if rTMS can reduce cocaine craving and use, and also affect several mood, behavioral and cognitive alterations associated with prolonged cocaine use.

Eligibility: Healthy, right-handed adults ages 18-65 who do have cocaine use disorder (moderate to severe).

Design: This is a randomized, double-blind, sham-controlled study. The study includes three phases: 1) a rTMS continued treatment phase; a rTMS follow-up; and a no rTMS follow-up.

Prior to participating, participants will be screened with:

* Questionnaires
* Medical history
* Physical exam
* Urine tests
* MRI (structural)

After being enrolled, baseline behavioral and imaging data will be collected. In particular, participants will undergo:

* Questionnaires
* Functional MRI

During the continued rTMS phase, participants with cocaine use disorder will be randomized to receive real or fake rTMS. Repetitive TMS will be delivered during 10 outpatient treatment days, over 2 weeks (5 days/week). Following this phase, subjects will have 12 follow-up visits (once/weekly), during which they will receive rTMS, and behavioral and imaging assessments will be performed. At the end of the rTMS follow up period, participants will further receive 3 follow up visits (once a month), during which rTMS will not be performed, but behavioral data will be collected.

Treatment includes:

* rTMS: A coil is placed on the head. A brief electrical current passes through the coil. At each visit, participants will receive two rTMS sessions, with a 1hr interval between sessions. At the beginning of each rTMS session, they view cocaine-related images for few minutes.
* MRIs at baseline and at follow-up visit #12: Participants lie on a table that slides into a cylinder that takes pictures of the brain. They respond to images while in the scanner.
* Repeat of screening tests and questionnaires
* Urine toxicological screen

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) has been shown to reduce craving in cocaine addicts. However, the efficacy of rTMS in treating cocaine addiction has not been evaluated in double-blind, sham-controlled studies and also, we lack a full characterization of rTMS effects on other important aspects, including effects on mood, cognition and changes in brain function. The purpose of this study is to investigate the effects of repetitive Transcranial Magnetic Stimulation (rTMS) at 15 Hz frequency on the left dorsolateral prefrontal cortex in cocaine dependent patients and to examine possible changes in mood, cognition, and brain activity and functional connectivity associated with this intervention. For this purpose, the investigators will recruit cocaine dependent patients. After screening and informed consent, participants will undergo active or sham rTMS for two consecutive weeks (twice a day) during the continued treatment phase, and a maintenance intervention (twice a week for 3 months), during the rTMs follow-up phase. Following this phase, participants will be followed for further 3 months, during which no rTMS will be delivered but clinical and imaging data will be collected. The investigators will also measure clinical, cognitive and brain structural and functional connectivity to assess changes related to the intervention in the short and long term (measurements at: baseline, 2 weeks, 3 months, 6 months).

Procedure: The project consists of: Screening Visit (baseline), Part 1 (continued treatment phase), Part 2 (3 months- rTMS follow-up), Part 3 (3 months follow-up without rTMS). First, there will be a screening visit, where a clinical interview will be conducted and questionnaires and tests will be administered to identify study participants who meet the inclusion and exclusion criteria. Baseline clinical, cognitive and neuroimaging data will be acquired. The neuroimaging data will be exploratory, to be associated with the outcome measures. In Part 1, all participants will be randomly assigned to one of the two treatment arms with rTMS (15Hz, 15Hz-Sham). Participants will receive 2 sessions of rTMS (active or sham), twice per day for 10 consecutive days, for a total of 20 rTMS sessions. Following this, the investigators will evaluate the acute effect of treatment on cocaine craving and consumption, mood and cognition. Also, they will collect exploratory neuroimaging data (functional MRI and resting state functional connectivity). In Part 2 of the study, all participants will continue the assigned treatment arm with rTMS (15Hz, 15Hz-Sham) for three months. Participants will receive 2 sessions of rTMS (active or sham) once per week; clinical and cognitive data will be acquired once per month. The investigators will evaluate the effect of treatment on cocaine craving and consumption, mood and cognition. Also, they will collect exploratory neuroimaging data (functional MRI and resting state functional connectivity). In Part 3 of the study, participants will not receive any rTMS session. Clinical and cognitive data will be acquired once per month for three months. The investigators will evaluate the long-term effect of treatment on cocaine craving and consumption, mood and cognition.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of cocaine use disorder (from moderate to severe), based on the Diagnostic and Statistical Manual of Mental Disorder - Fifth Edition (DSM-5);
2. Abstinence from cocaine for at least 48 hrs.

Exclusion Criteria:

1. Current DSM-5 diagnosis of substance and/or alcohol use disorders other than nicotine;
2. Current DSM-5 diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder;
3. Use in the past 4 weeks of any medication with known pro-convulsant action; or current regular use of any psychotropic medications (benzodiazepines, antipsychotic medications, tricyclic antidepressants, anti-epileptics, mood stabilizers);
4. Any history of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes;
5. Any personal or family history (1st degree relatives) of seizures other than febrile childhood seizures;
6. Any psychiatric, medical or social condition whether or not listed above, due to which, in the judgment of the PI and after any consults if indicated, participation in the study is not in the best interest of the patient;
7. For female patients: Pregnancy/breastfeeding.
8. Subjects who have contraindications to MRI. Some of the exclusions are:

   1. Have non-MRI compatible metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or ferromagnetic fragments in the eye or oral cavity as these make having an MRI unsafe.
   2. Unable to lie flat on the back for the expected length of the experiment (50 minutes).
   3. Have an abnormality on the brain imaging or neurologic examination not related to the diagnosis.
   4. Uncomfortable being in a small space for the expected length of the experiment (50 minutes).
   5. Non-removable body piercing or tattoo posing MRI risk
   6. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Brief Version of Cocaine Craving Questionnaire (Brief-CCQ) Total score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  Brief Version of Cocaine Craving Questionnaire (Brief-CCQ) is a 10-item scale that evaluates craving for cocaine. Each Brief-CCQ item is rated on a 1 to 7 scale. The Brief-CCQ Total score ranges from 10 (min) to 70 (max). Higher Brief-CCQ scores indicate higher cocaine craving levels.
Change in cocaine consumption as assessed by Timeline Follow Back (TLFB) | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months, 12 months
  Cocaine consumption will be assessed using the TimeLine Follow Back (TLFB). TLFB is an interview-based assessment. Using a calendar, participants are guided through the process of recalling and reporting daily substance consumption. TLFB provides measures of cocaine consumption per week, cocaine consuming days per week, heavy cocaine consuming days per week.
Change in cocaine consumption as assessed by Urine Drug Screen (UDS) | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months, 12 months
  Cocaine consumption will be evaluated by Urine Drug Screen (UDS). Urine Drug Screen is a painless test to evaluate the presence of cocaine and other substances of abuse in urine samples. Quantitative analyses are not performed. Test may be positive or negative for the presence of cocaine and other substances.

SECONDARY OUTCOMES:
Changes in 90 Symptom Checklist (SCL-90) Global indices | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Symptom Checklist-90 (SCL-90) is a 90-item self-report psychometric instrument. It takes 12-15 minutes to administer. Each item is rated on a scale from 0 (not at all) to 5 (extremely). The global Indices include the General Severity Index (GSI), which is the average rating to all 90 items, the Positive Symptom Total (PST), which is the number of symptoms complained (items scored above zero), and the Positive Symptom Distress Index (PSDI), which is the average rating given to complained symptoms (items scored above zero).
Changes in Montgomery-Asberg Depression Scale (MADRS) Total Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The MADRS is a 10-item scale that evaluates the core symptoms and cognitive features of clinical depression. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Changes in Hamilton Rating Scale for Anxiety (HAM-A) Total Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The HAM-A is a 14-item scale that assesses anxiety symptoms of anxiety such as "anxious mood", "tension" or "fears". Each item is scored on a 5-point scale, ranging from 0 (not present) to 4 (severe). Sum the scores from all 14 parameters gives the HAM-A Total Score which may range from 0 (min) to 56 (max).
Changes in the Frontal Assessment Battery (FAB) Total Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  Frontal Assessment Battery (FAB) is a short neuropsychological tool aimed at assessing executive functions. The FAB consists of six subtests, each exploring functions related to the frontal lobes: conceptualization (by means of a similarities task), mental flexibility (by means of a phonological fluency task), motor programming (by means of Luria's motor series), sensitivity to interference (by means of a conflicting instructions task), inhibitory control (by means of a go-no-go task), and environmental autonomy (by means of evaluation of prehension behavior). Each subtest score may range from 0 (min) to 3 (max); total score is from 0 (min) to 18 (max). Higher scores indicate better performance.
Changes in Eriksen Flanker Test | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Eriksen Flanker Task is a set of response inhibition tests used to assess the ability to suppress responses that are inappropriate in a particular context. The target is flanked by non-target stimuli which correspond either to the same directional response as the target (congruent flankers), to the opposite response (incongruent flankers), or to neither (neutral flankers). A directional response (usually left or right) is assigned to a central target stimulus. Each task begin with a short instruction phase followed by 20 practice trials and 100 experimental trials. The stimuli are displayed for 1500 msec. The measures of performance in each condition is the median reaction time (RT) for correct trials and the proportion of errors.
Changes in the Iowa Gambling Task (IGT) Performance | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Iowa Gambling Task is a computerized card game commonly used to measure risky decision making tendencies and sensitivity to reward and loss. Performance is calculated on the total net score results from the subtraction of the disadvantageous deck choices from the advantageous deck choices during the entire test ([C'+D']-[A'+B']).
Changes in Snaith Hamilton Pleasure Scale (SHAPS) Total Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Snaith Hamilton Pleasure Scale (SHAPS) is a 14-item self-report scale designed to measure hedonic-tone/anhedonia. Each item is scored on a 4-point scale, ranging from 0 (not at all) to 3 (extremely). Sum the scores from all 14 parameters gives the SHAPS Total Score which may range from 0 (min) to 42 (max).
Changes in Temporal experience of Pleasure Scale (TEPS) Total Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Temporal experience of Pleasure Scale (TEPS) is a 18-item self-report scale designed to evaluate individual trait dispositions in anticipatory and consummatory pleasure experiences. Each item is scored on a 6-point scale, ranging from 1 (extremely false) to 6 (extremely true). Sum the scores from all 20 parameters gives the TEPS Total Score which may range from 20 (min) to 108 (max).
Changes in Profile of Mood States (POMS), Total Mood Disturbance Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The profile of mood state (POMS) is a questionnaire designed to measure present mood state by a list of adjectives on a 5-point Likert scale (0 = not at all; 4 = Extremely) and measures six dimensions of affect, including tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. The measure has been shown to produce reliable and valid profiles of mood state. A Total Mood Disturbance Score may be calculated by adding the scores for Tension, Depression, Anger, Fatigue and Confusion and then subtracting the score for Vigour.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo di Giannantonio, MD, Principal Investigator — Department of Neuroscience, Imaging and Clinical Sciences (ITAB) - University G. d'Annunzio - Chieti (Italy)
Locations (2):
- Italy (2):
  - Department of Neuroscience, Imaging and Clinical Sciences, Chieti
  - La Promessa ONLUS, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinotti G, Pettorruso M, Montemitro C, Spagnolo PA, Acuti Martellucci C, Di Carlo F, Fanella F, di Giannantonio M; Brainswitch Study Group. Repetitive transcranial magnetic stimulation in treatment-seeking subjects with cocaine use disorder: A randomized, double-blind, sham-controlled trial. Prog Neuropsychopharmacol Biol Psychiatry. 2022 Jun 8;116:110513. doi: 10.1016/j.pnpbp.2022.110513. Epub 2022 Jan 22. PMID 35074451
- [Derived] Pettorruso M, Spagnolo PA, Leggio L, Janiri L, Di Giannantonio M, Gallimberti L, Bonci A, Martinotti G. Repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex may improve symptoms of anhedonia in individuals with cocaine use disorder: A pilot study. Brain Stimul. 2018 Sep-Oct;11(5):1195-1197. doi: 10.1016/j.brs.2018.06.001. Epub 2018 Jun 5. No abstract available. PMID 29885861

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT03333460/Prot_SAP_000.pdf